CLINICAL TRIAL: NCT05388643
Title: Early Detection of Gestational Diabetes Mellitus in Pregnancy: A Randomized Trial
Brief Title: Early Detection of Gestational Diabetes Mellitus in Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Gianna Wilkie, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: STUDY00002047; K23HD111526 (NIH)
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy; Pregnancy, High Risk
Keywords: Pregnancy; Gestational Diabetes; Screening; Maternal Outcomes; Neonatal Outcomes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, randomized study evaluating an early screening protocol for identifying women at high risk for developing GDM to the routine standard of care for GDM screening.
Who Masked: Outcomes Assessor
Masking Description: Those assessing the outcomes from the medical chart will be blinded to the randomization process and the assigned study arm. Patients, the primary investigator, and their care providers will be aware of their treatment status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Enhanced First Trimester GDM Screening (Experimental): Women who are randomly assigned to this condition will be required to have early glucose screening with a prediction model composed of additional clinical risk factors and serum biomarkers (triglycerides, PAPP-A, and lipocalin-2) with their initial prenatal laboratory assessment.
  Interventions: Diagnostic Test: Enhanced First Trimester GDM Screening
- Standard of Care GDM Screening (Active Comparator): Women who will be randomized to the comparison condition of usual standard of care will undergo routine standard of care. The standard of care will consist of routine screening for diabetes in pregnancy between 24 to 28 weeks of gestation via the two-step screening method with possible early screening with either plasma fasting glucose, oral glucose tolerance test, or hemoglobin A1c at the providers discretion to represent true clinical practice.
  Interventions: Diagnostic Test: Routine Gestational Diabetes Screening

INTERVENTIONS:
Diagnostic Test: Enhanced First Trimester GDM Screening — Women who are randomly assigned to this condition will be required to have early glucose screening with a prediction model composed of additional clinical risk factors and serum biomarkers (triglycerides, PAPP-A, and lipocalin-2) with their initial prenatal laboratory assessment.
  Arms: Enhanced First Trimester GDM Screening
Diagnostic Test: Routine Gestational Diabetes Screening — Women who will be randomized to the comparison condition of usual standard of care will undergo routine standard of care. The standard of care will consist of routine screening for diabetes in pregnancy between 24 to 28 weeks of gestation via the two-step screening method with possible early screening with either plasma fasting glucose, oral glucose tolerance test, or hemoglobin A1c at the providers discretion to represent true clinical practice.
  Other Names: Third Trimester Screening
  Arms: Standard of Care GDM Screening

SUMMARY:
The purpose of this study is to develop an implementation protocol and test the feasibility and acceptability of a first trimester screening protocol for the early detection of gestational diabetes mellitus (GDM).

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is an important contributor to both maternal and neonatal morbidity and mortality in pregnancy. GDM has lifelong complications including an increased risk of developing type 2 diabetes mellitus and cardiovascular disease for women, and their offspring are at higher risk of being obese and also having diabetes in childhood and adolescence. Approximately 1 in 8 pregnancies is impacted by gestational diabetes mellitus worldwide. First trimester GDM screening is varied due to conflicting national guidelines, and the best strategy is unknown. The goal of the proposed research is to develop an implementation protocol and test the feasibility and acceptability of a first trimester screening protocol for the early detection of GDM. The investigators will utilize a pilot randomized controlled trial to recruit 80 high-risk pregnant women in the first trimester, of whom half will receive protocolized early GDM screening with serum biomarkers before 12 weeks and the remaining half will receive the current standard of care with screening between 24 and 28 weeks of gestation with possible early screening based on provider discretion.

ELIGIBILITY:
Inclusion Criteria:

* 1) age greater than or equal to 18 years old,
* 2) singleton gestation less than or equal to 12 weeks at initial obstetric visit,
* 3) receiving prenatal care at UMMHC and plans to deliver at UMMHC,
* 4) able and willing to provide informed consent,
* 5) English or Spanish speaking, and
* 6) are at high risk for developing GDM by ACOG clinical risk factor guidelines.

Exclusion Criteria:

* 1) known diagnosis of pre-existing pregestational diabetes,
* 2) plan to receive prenatal care or deliver outside of UMMHC,
* 3) inability to complete oral glucose tolerance test (e.g. gastric bypass surgery history, gastric dumping syndrome history, vomiting of oral glucose tolerance test), or
* 4) systemic steroid use.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Gestational Diabetes Mellitus | In pregnancy (24-28 weeks gestation)
  Confirmed diagnosis of GDM based on 3 hour 100 gram glucose tolerance test

SECONDARY OUTCOMES:
Mode of Delivery | At Birth
  Mode of delivery (Vaginal versus Cesarean delivery)
Neonatal Birthweight | At Birth
  Neonatal Birthweight
Number of Participants with Shoulder Dystocia | At Birth
  Number of Participants with Shoulder Dystocia
Number of participants with brachial plexus injury | At Birth
  Number of participants with brachial plexus injury
APGAR Score | At Birth
  APGAR Score (range 0 to 10, with 10 being the best)
Neonatal Intensive Care Unit Admission | At delivery and within first 2 days of life
  Admission to Level 2 or greater neonatal ICU and length of stay
Gestational Age at Delivery | At Birth
  Gestational Age at Delivery
Patient Satisfaction with Diabetes Screening Method | Postpartum day 1 after birth
  This will be assessed by the Patient Satisfaction Survey questionnaire, which is scored out of 30, with 30 being the highest score)

CONTACTS AND LOCATIONS:
Overall Officials: Gianna Wilkie, MD, Principal Investigator — University of Massachusetts Chan Medical School
Locations (1):
- University of Massachusetts Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sweeting AN, Wong J, Appelblom H, Ross GP, Kouru H, Williams PF, Sairanen M, Hyett JA. A Novel Early Pregnancy Risk Prediction Model for Gestational Diabetes Mellitus. Fetal Diagn Ther. 2019;45(2):76-84. doi: 10.1159/000486853. Epub 2018 Jun 13. PMID 29898442
- [Result] Nanda S, Savvidou M, Syngelaki A, Akolekar R, Nicolaides KH. Prediction of gestational diabetes mellitus by maternal factors and biomarkers at 11 to 13 weeks. Prenat Diagn. 2011 Feb;31(2):135-41. doi: 10.1002/pd.2636. Epub 2010 Dec 28. PMID 21268030